CLINICAL TRIAL: NCT01831219
Title: A Follow-Up Study of Subjects Enrolled in the Pin-Based (IDE G920035) and Pinless (IDE G000071) ROBODOC® Surgical System Clinical Trial
Brief Title: ROBODOC® Clinical Trials: Long-Term Follow-Up
Status: Completed | Type: Observational
Sponsor: Curexo Technology Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-PROTO-01
Record Dates: First submitted 2013-04-09; First posted 2013-04-15 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; arthroplasty; hip arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ROBODOC: The ROBODOC group received total hip arthroplasty using the ROBODOC Surgical system for preparation of the femoral canal for a femoral stem implant.
- Conventional: The conventional group received total hip arthroplasty using the conventional manual tools including a broach to prepare the femoral cavity for femoral stem replacement.

SUMMARY:
This is a follow-up study looking at the and long-term results of two methods of preparing the thigh bone to receive an implant during hip replacement surgery. For one group of patients in the original study, the surgeon used a cutting tool called a broach and a special hammer on patients who had standard hip replacement operations. For the other patients, the surgeon used a surgical robot which was equipped with a cutting tool, like a drill, to prepare the thigh bone. The purpose of this study is to collect additional information confirming that the surgical robot is safe and effective when used as recommended. Only patients who were enrolled in the original clinical trials are eligible for this study.

DETAILED DESCRIPTION:
A. Description This study is a follow-up study looking at mid- and long-term outcomes for participants in the IDE G920035 and IDE G000071 Clinical Trials. The IDE G920035 was a randomized, controlled trial with a 1:1 ROBODOC:control randomization. The IDE G000071 was a randomized, controlled trial with a 3:1 ROBODOC:control randomization.

B. Selection Criteria Only subjects who were originally enrolled in the IDE G920035 and IDE G000071 Clinical Trials are eligible to participate in this study. Subjects selected for this study will have completed a minimum of the 3 month follow-up requirements of the IDE G920035 and IDE G000071 Clinical Trials. Enrolled subjects must be willing to give a relevant medical history, undergo a focused physical examination of their operative hip(s), have an AP and lateral x-ray taken of their operative hip(s) and complete the Harris Hip Score, SF-12, UCLA Activity Score, VAS pain self-assessment, and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaires.

The study subject may be reimbursed for reasonable travel expenses associated with their participation in the study. All requests for reimbursement must be pre-approved by Curexo Technology Corporation.

C. Data Collection Subjects participating in this study will be asked to visit the study site to undergo a physical examination of their operative hip(s). During this visit, they will be asked to give a relevant medical history, have AP and lateral radiographs taken of their operative hip(s), and complete the Harris Hip Score, SF-12, UCLA Activity Score, VAS pain self-assessment, and WOMAC questionnaires.

If the subject has obtained AP and lateral radiographs within the last year, these can be used instead of requiring them to obtain new radiographs specifically for this study.

If the subject is unable or unwilling to come in for the examination, they will be asked to fill out the Harris Hip Score, SF-12, UCLA Activity Score, VAS pain self-assessment, and WOMAC questionnaires via mail or over the phone with the Study Nurse/Coordinator. Additionally, they will be asked to obtain current AP and lateral radiographs taken of their operative hip(s) with their current orthopaedic surgeon to be transferred to the study site.

D. Blinding An independent radiologist or orthopaedic surgeon, experienced in reading hip x-rays, who is blinded to the original randomly assigned study group, will read the follow-up x-rays taken on subjects enrolled in this study.

E. Randomization There will be no further randomization of subjects in this study. Prior subject records will determine the original study group (ROBODOC or manual control) to which the subject was randomly assigned in IDE G920035 or IDE G000071.

F. Baseline Measurements No baseline measurements will be collected for this follow-up study. G. Power and Sample Size The sample size will be determined by the number of qualifying subjects from the IDE G920035 and IDE G000071 Clinical Trials who can be located and who agree to participate in this follow-up study. We anticipate approximately 20 patients from IDE G920035 and 30 patients from IDE G000071 to agree to study participation. This sample size will provide 82% power (α = 0.05, 2-tailed) to detect a 20% (5 versus 2.5, pooled SD = 3.0) difference between the ROBODOC and control groups on the VAS at the last available follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects included in this study will have completed the follow-up requirements of the IDE G920035 or the IDE G000071 Clinical Trial;
* Subjects must be willing to give a relevant medical history, undergo a focused physical examination of their operative hip(s) and have an AP and lateral x-ray taken of their operative hip(s);
* Subjects must be willing to complete the Harris Hip Score, SF-12, WOMAC, UCLA Activity Score, and VAS pain self-assessment questionnaires; and
* Subjects must be willing to sign an informed consent document.

Exclusion Criteria:

* There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects included in this study will have been enrolled in either the IDE G920035 or the IDE G000071 Clinical Trial and will have completed the follow-up requirements to those trials.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2013-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William L Bargar, MD, Principal Investigator — Department of Orthopaedics, University of California at Davis
Locations (1):
- Sutter Institute for Medical Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bargar WL, Bauer A, Borner M. Primary and revision total hip replacement using the Robodoc system. Clin Orthop Relat Res. 1998 Sep;(354):82-91. doi: 10.1097/00003086-199809000-00011. PMID 9755767

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ROBODOC | Conventional
Started | 73 | 45
Completed | 40 | 21
Not Completed | 33 | 24

BASELINE CHARACTERISTICS:
Population: Patients enrolled in IDE G920035 trial or IDE G000071 trial and underwent total hip arthroplasty using either the ROBODOC Surgical Assistant System or a manual technique.
Groups:
- Total: Total of all reporting groups
Arm/Group | ROBODOC | Conventional | Total
Number analyzed (Participants) | 73 | 45 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 73 | 45 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (8.2) | 72.8 (7.6) | 73.5 (7.7)
Gender [Count of Participants; unit: Participants]
  Female | NA — The gender breakdown of the original IDE was collected but it is unavailable, because the data has been lost. | NA — The gender breakdown of the original IDE was collected but it is unavailable, because the data has been lost. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — The gender breakdown of the original IDE was collected but it is unavailable, because the data has been lost. | NA — The gender breakdown of the original IDE was collected but it is unavailable, because the data has been lost. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 73 | 45 | 118

OUTCOME MEASURES:

1. Primary Outcome: Presence of Osteolysis
Description: Presence of osteolysis determined by looking at patient x-rays as described by Gruen et al and Johnson et al.
Time Frame: 14 months
Measure: Number; unit: Hips
Units Other Than Participants: Hips
Arm/Group | ROBODOC | Conventional
Number analyzed (Participants) | 40 | 21
Number analyzed (Hips) | 45 | 22
Hips | 2 | 2

2. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index
Description: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) will be used to measure clinical outcome. The WOMAC total score ranges 96 (best) to 0 (worst). The WOMAC pain score ranges 0-20, the stiffness score ranges 0-8, and functional limitation score ranges 0-68.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Arm/Group | ROBODOC | Conventional
Number analyzed (Participants) | 40 | 21
Number analyzed (Hips) | 45 | 22
units on a scale | 8.44 (11.48) | 11.32 (11.92)

3. Secondary Outcome: Harris Hip Score
Description: The Harris Hip Score will be measured to determine clinical outcome. The Harris Hip total score ranges 100 (best) to 0 (worst) and it is computed by the sum of the pain score (0-44 points), function (, 0-47 points), absence of deformity (4 points), and range of motion (5 points).
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Arm/Group | ROBODOC | Conventional
Number analyzed (Participants) | 40 | 21
Number analyzed (Hips) | 45 | 22
units on a scale | 93.49 (8.77) | 89.5 (12.03)

4. Secondary Outcome: Health Status Questionnaire-12
Description: The Health Status Questionnaire-12 (HSQ-12) will be used to measure clinical outcome. HSQ-12 total score ranges from 0 (worst) to 800 (best).
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Arm/Group | ROBODOC | Conventional
Number analyzed (Participants) | 40 | 21
Number analyzed (Hips) | 45 | 22
units on a scale | 683.52 (113.09) | 637.16 (104.53)

5. Secondary Outcome: UCLA Activity Score
Description: The UCLA Activity Score will be used to measure clinical outcome. The UCLA Activity Score ranges 10 (best) to 0 (worst).
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Arm/Group | ROBODOC | Conventional
Number analyzed (Participants) | 40 | 21
Number analyzed (Hips) | 45 | 22
units on a scale | 6.09 (8.44) | 5.71 (1.45)

6. Secondary Outcome: Visual Analog Pain Score
Description: The Visual Analog Scale pain questionnaire will be used to measure clinical outcome. The pain VAS is a continuous scale which range from 0 (no pain) to 100 [100-mm scale] ("worst imaginable pain" ).
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Arm/Group | ROBODOC | Conventional
Number analyzed (Participants) | 40 | 21
Number analyzed (Hips) | 45 | 22
units on a scale | 4.69 (10.15) | 6.42 (10.89)

7. Other Pre Specified Outcome: Number of Operated Hips That Required Revision/Reoperation
Description: Implant survivorship will be determined from the medical history CRF by comparing the percentage of ROBODOC and manual control subjects who have required revision or re-operation THA procedures on the hip in question since their original study procedure which took place 7-20 years previously.
Time Frame: At follow-up visit (7-20 years post-operatively)
Measure: Number; unit: Hips
Units Other Than Participants: Hips
Arm/Group | ROBODOC | Conventional
Number analyzed (Participants) | 40 | 21
Number analyzed (Hips) | 45 | 22
Hips | 1 | 1

ADVERSE EVENTS:
Time Frame: 2 years, 2 months
Groups:
- ROBODOC: The ROBODOC group received total hip arthroplasty using the ROBODOC Surgical sys...
Arm/Group | ROBODOC | Conventional
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/21
Other Adverse Events (participants affected / at risk) | 0/40 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No